CLINICAL TRIAL: NCT06649461
Title: Splint with Ozone Injection for Mild and Moderate Carpal Tunnel: an Electrodiagnostic Study
Brief Title: Efficacy of Ozone Therapy and Splint in Carpal Tunnel Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Emine Cihan, Assist. Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/10.6
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: splint; ozone therapy; rehabilitation
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ozone injections (Experimental)
  Interventions: Procedure: ozone injections; Other: Splint
- splint (Active Comparator)
  Interventions: Other: Splint

INTERVENTIONS:
Procedure: ozone injections — Ozone injections (5 mL/10 μg/dL) were administered under aseptic conditions, with the wrist fixed in dorsiflexion, and with the insulin injector, a 23-gauge needle was inserted between the palmaris longus and flexor carpi radialis muscles at a 45-degree angle from the palmar distal line (Salutem/19147884379).
  Arms: ozone injections
Other: Splint — hand splint for night

SUMMARY:
This study will investigate the effectiveness of repeated ozone therapy combined with splint therapy for carpal tunnel syndrome (CTS).CTS patients will be split into two groups: ozone plus splint and splint only. Both groups will use wrist splints for 3 weeks, with the ozone+splint group receiving weekly ozone injections for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* being 18-65 years, with mil-modarete CTS, symptoms continued for at least 3 months

Exclusion Criteria:

* hand edema or prior injections, thenar atrophy, prior CTS surgery, severe EMG results, recent physical therapy, steroids, or platelet-rich plasma for CTS in the past year, and conditions causing secondary CTS (e.g., thyroid disorders, diabetes, pregnancy, rheumatoid arthritis, Dupuytren's contracture, inflammatory arthritis, connective tissue diseases). Also excluded: neck or arm pain conditions (e.g., cervical disc herniation, wrist fracture, proximal upper extremity entrapment neuropathy, polyneuropathy, peripheral nerve damage, fibromyalgia), history of G6PD deficiency, uncontrolled hyperthyroidism, thrombocytopenia, and contraindications to general ozone therapy (e.g., ACE inhibitors for severe cardiovascular instability).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-10-29 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire | 10 minutes
  As the score obtained from the survey increases, the improvement increases.
visual analog scale | 1 minute
  As the score approaches 10, the intensity of pain felt increases.
electromyography (EMG) | 10 minutes
  In the electrophysiological examination, median sensory nerve conduction studies and median motor nerve conduction studies will be measured. Median motor nerve latency, median motor nerve conduction velocity, and compound muscle action potential amplitude will be measured and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No